CLINICAL TRIAL: NCT06597760
Title: A Clinical Study to Evaluate the Effect of Enlicitide on the Pharmacokinetics of Digoxin in Healthy Adult Participants
Brief Title: A Clinical Study to Assess the Effect of Enlicitide on How the Body Processes Digoxin in Healthy Adult Participants (MK-0616-031)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0616-031; MK-0616-031 (Other: MSD); CA41814 (Other: Celerion)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: 0.25mg Digoxin-->0.25mg Digoxin plus 20mg enlicitide/180mg Sodium Caprate (Experimental): Participants will receive 1 tablet of 0.25mg Digoxin on Day 1 of period 1 and 1 tablet of 0.25mg Digoxin coadministered with 1 tablet of 20 mg enlicitide/180 mg sodium caprate on Day 1 of Period 2.
  Interventions: Drug: Enlicitide; Drug: Digoxin
- Sequence 2: 0.25mg Digoxin plus 20mg enlicitide/180mg Sodium Caprate-->0.25mg Digoxin (Experimental): Participants will receive 1 tablet of 0.25mg Digoxin coadministered with 1 tablet of 20 mg enlicitide/180 mg sodium caprate on Day 1 of Period 1 and will receive 1 tablet of 0.25mg Digoxin on Day 1 of period 2.
  Interventions: Drug: Enlicitide; Drug: Digoxin

INTERVENTIONS:
Drug: Enlicitide — Participants will receive 20 mg enlicitide/180 mg sodium caprate coadministered with 0.25mg Digoxin orally on Day 1, Period 2 in Arm A and on Day 1 Period 1 in Arm B.
  Other Names: enlicitide decanoate; MK-0616/sodium caprate
Drug: Digoxin — Participants will receive 0.25 mg digoxin orally on Day 1 Period 1 in Arm A and Day 1 Period 2 in Arm B. They also receive Digoxin orally on Day 1, Period 2 in Arm A and on Day 1 Period 1 in Arm B coadministered with oral 20 mg enlicitide/180 mg sodium caprate.

SUMMARY:
Researchers have designed a new study medicine called enlicitide decanoate as a new way to lower the amount of low-density lipoprotein cholesterol (LDL-C) in a person's blood. Enlicitide decanoate will be called "enlicitide" from this point forward.

The purpose of this study is to learn the effect of this new study medicine enlicitide on digoxin (medicine used in heart disease) over time (a pharmacokinetic or PK study). Researchers will compare what happens to digoxin in the body over time when it is given with this new study medicine enlicitide in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has a body mass index (BMI) ≥18 and ≤32 kg/m^2, inclusive

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant psychiatric, immunological, gastrointestinal, cardiovascular abnormalities or diseases.
* Has a history of cancer.
* Has positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at the screening visit.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) for Digoxin in Plasma | At designated timepoints (up to 5 days)
  AUC0-inf is the area under the plasma concentration versus time curve (AUC) for digoxin, from time zero (pre-dose) to extrapolated infinite time.

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUC0-last) for Digoxin in Plasma | At designated timepoints (up to 5 days)
  Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration is at or above the lower limit of quantification (LLQ).
Cmax (Maximum Concentration) for Digoxin in Plasma | At designated timepoints (up to 5 days)
  Blood samples will be collected at at designated timepoints (up to 5 days) post-dose to determine the Cmax of Digoxin.
Tmax (Time to Maximum Concentration) for Digoxin in Plasma | At designated timepoints (up to 5 days)
  The time to reach Cmax (Tmax) is determined. Blood samples will be collected at designated timepoints (up to 5 days) post-dose to determine the maximum concentration (Cmax) of digoxin.
Terminal half life (T½) for Digoxin in Plasma | At designated timepoints (up to 5 days)
  T1/2 is defined as the time taken for the plasma concentration or the amount of digoxin in the body to be reduced by half.
Apparent Clearance (CL/F) for Digoxin in Plasma | At designated timepoints (up to 5 days)
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Apparent Volume of Distribution During Terminal Phase (Vz/F) for Digoxin in Plasma | At designated timepoints (up to 5 days)
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/f after oral dose of digoxin is influenced by the fraction absorbed.
Number of Participants With Treatment Emergent Adverse Events (TEAEs): | Up to ~ 28 days.
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs are defined as all AEs that occurred at or after the first dose of the investigational product and through the last follow-up date.
Number of Participants With Clinical Laboratory Abnormalities | Up to ~ 28 days
  Clinical laboratory test include serum chemistry, hematology and urinalysis. Clinical laboratory abnormalities were recorded and reported as TEAE. TEAEs are defined as all AEs that occurred at or after the first dose of the investigational product or device implant surgery (whichever occurred earlier) and through the last follow-up date.
Standard and Orthostatic Vital Signs | Up to ~ 28 days
  Single measurements of body temperature, respiratory rate, blood pressure, and heart rate, and triplicate measurements of blood pressure and heart rate will be measured. Orthostatic vital signs (i.e., heart rate and blood pressure) will be measured, Measurements will be collected with participants in a semi-recumbent position and then collected when in a standing position.
12-lead Electrocardiogram (ECGs) | Up to ~ 28days
  Single and triplicate 12-lead ECGs will be performed. Triplicate 12-lead ECGs will be performed within an approximately 6-minute time window. ECGs will be performed with participants in a supine position for at least 5 minutes. In each period, triplicate ECGs will be measured within 3 hours prior to dosing. When scheduled post dose, single ECGs will be performed within ±20 minutes of the scheduled time point.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com